CLINICAL TRIAL: NCT02679534
Title: The Effectiveness of Hand Massage on the Pain of Cardiac Surgery Critically Ill- A Randomized Controlled Trial
Brief Title: The Effectiveness of Hand Massage on the Pain of Cardiac Surgery Critically Ill
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Céline Gélinas, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-186
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Pain
Keywords: pain; thoracic surgery; massage
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- hand massage (Experimental): Patients will receive a 20 minute hand massage by a trained nurse in addition to the standard ICU care. Before administering the massage, a favorable environment will be created that promotes calmness such as dampening the light, reducing the alarm intensity, closing the curtains and the door and posting the notice "do not disturb", and a comfortable positioning of the patient will be ensured. The interventionist will hold each hand for 5-10 seconds, and apply 5-10 ml of unscented hypoallergenic cream to both hands and wrists. Then, she will perform massage using moderate pressure, and the stroking and kneading techniques during ten minutes on the palm and back of each hand.
  Interventions: Other: hand massage; Other: application of unscented hypoallergenic cream; Other: environmental adjustments
- hand holding (Active Comparator): The active control group will receive hand holding by the same trained nurse in addition to standard ICU care. The same hand hygiene and environmental adjustments will be made as for those receiving massage. Patients will have their hands held for 5-10 seconds and unscented hypoallergenic cream applied to both hands. Then, the interventionist will hold each of the patients' hand in her hand for ten minutes without performing any tissue manipulation. The hand holding procedure will last for a total of 20 minutes.
  Interventions: Other: hand holding; Other: application of unscented hypoallergenic cream; Other: environmental adjustments
- rest group (Other): The passive control group will have a 20 minutes rest period including the same environmental adjustments as the massage and hand holding groups in addition to the standard care administered in the ICU. The standard care includes the pharmacological and non-pharmacological treatments used to promote recovery and symptom relief. In the study ICU, cardiac surgery patients are automatically prescribed a pain management protocol that includes the regular administration of morphine, unless extraordinary patient circumstances require different prescriptions. Patients might equally receive breakthrough doses of analgesia in addition to regular opioids. Of the existing non-pharmacological interventions, repositioning and back rubs are commonly employed in the study ICU to provide patient comfort.
  Interventions: Other: environmental adjustments

INTERVENTIONS:
Other: hand massage
  Arms: hand massage
Other: hand holding
  Arms: hand holding
Other: application of unscented hypoallergenic cream
  Arms: hand holding; hand massage
Other: environmental adjustments

SUMMARY:
Postoperative pain is a common phenomenon in the intensive care unit (ICU) despite the multitude of efforts dedicated to promote its effective relief. Mounting evidence shows that cardiac surgery ICU patients experience moderate to severe pain reaching proportions as high as 74% despite the use of analgesics. The highest pain intensity is experienced in the first 24 hours post surgery when patients are still in the ICU, and represents a strong predictor for the presence and severity of persistent postoperative pain. To maximize pain relief, massage has been suggested in the recent clinical practice guidelines of the Society of Critical-Care Medicine as a complementary non-pharmacological therapy in the ICU given its opioid-sparing and analgesia-enhancing potential. Some randomized controlled trials showed promising pain relief effects of massage when administered to cardiac surgery patients in acute care units, however, its effects on pain relief while patients are still in the ICU and when pain severity is highest remain unknown.

This study aims to compare the effect of three 20-minute hand massage administrations within 24 hours postop on the pain intensity (primary outcome), pain unpleasantness, pain interference, muscle tension, anxiety and vital signs (blood pressure, heart and respiratory rates) of adult intensive care unit (ICU) patients post cardiac surgery versus hand holding (i.e., simple touch) and standard care. Other objectives are to describe the location and quality of pain of cardiac surgery ICU patients.

Hypothesis:

Patients receiving 3 hand massages within 24 hours postop will have lower pain intensity, unpleasantness and interference, muscle tension, anxiety and vital signs compared to patients receiving hand holding and to those in the standard care group.

ELIGIBILITY:
Inclusion Criteria:

* able to speak French or English
* elective cardiac surgery requiring sternal incision (e.g., coronary artery bypass graft, valve replacement)
* able to answer questions and self-report symptoms

Exclusion Criteria:

* previous cardiac surgery
* diagnostic of cognitive or psychiatric disorder
* pulmonary artery pressure >50 mmHg
* right ventricular failure
* systolic left ventricular dysfunction (ejection fraction 35% or less)
* body mass index > 30
* prolonged bleeding from the chest drainage tubes (i.e., >200 ml/h)
* having mechanical blood pressure support (e.g., intra-aortic balloon pump)
* receiving cardiac pacing with complete control of HR
* peripheral intravenous line in the hands
* suppurating/infective/inflammatory skin condition of the hands
* hypersensitivity to touch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
change in pain intensity from pre- to post-intervention as assessed using the 0-10 Numeric Rating Scale | before and immediately after each intervention within 24 hours postoperatively
  Pain intensity will be captured using the 0 to 10 Numeric Rating Scale score, and the analysis metric will be the change in pain intensity from baseline (pre-intervention) to immediately after each intervention. For each study group, means and standard deviations of patients' pain intensity levels will be reported.
  Change in pain intensity levels will be assessed for each of the three interventions administered within 24 hours postop.

SECONDARY OUTCOMES:
change in pain unpleasantness from pre- to post-intervention as assessed using the 0-10 Numeric Rating Scale | before and immediately after each intervention within 24 hours postop
change in muscle tension from pre- to post-intervention by performing passive flexion and extension of patient's arm, and scoring 0 (relaxed), 1 (tense) or 2 (very tense/rigid) | before and immediately after each intervention within 24 hours postop
  The muscle tension ordinal scale 0-2 is based on the muscle tension item of the Critical-Care Pain Observation Tool, a behavioral pain scale for the assessment of pain in the non-verbal critically ill.
change in anxiety from pre- to post-intervention as assessed using the 0-10 Numeric Rating Scale | before and immediately after each intervention within 24 hours postop
changes in 1-minute blood pressure average from pre- to post-intervention as assessed using a data collection computer connected to patient's bedside monitor | before and immediately after each intervention within 24 hours postop
changes in 1-minute heart rate average from pre- to post-intervention as assessed using a data collection computer connected to patient's bedside monitor | before and immediately after each intervention within 24 hours postop
changes in 1-minute respiratory rate average from pre- to post-intervention as assessed using a data collection computer connected to patient's bedside monitor | before and immediately after each intervention within 24 hours postop
pain interference as assessed using the Brief Pain Inventory | on the second and fourth postoperative days
change in pain intensity from post-intervention to 30 minutes later as assessed using the 0-10 Numeric Rating Scale (carry-over effect) | immediately after each intervention and 30 minutes later within 24 hours postop
change in pain unpleasantness from post-intervention to 30 minutes later as assessed using the 0-10 Numeric Rating Scale (carry-over effect) | immediately after each intervention and 30 minutes later within 24 hours postop
change in muscle tension from post-intervention to 30 minutes later by performing passive flexion and extension of patient's arm, and scoring 0 (relaxed), 1 (tense) or 2 (very tense/rigid) | immediately after each intervention and 30 minutes later within 24 hours postop
change in anxiety from post-intervention to 30 minutes later as assessed using the 0-10 Numeric Rating Scale (carry-over effect) | immediately after each intervention and 30 minutes later within 24 hours postop
changes in 1-minute blood pressure average from post-intervention to 30 minutes later as assessed using a data collection computer connected to patient's bedside monitor | immediately after each intervention and 30 minutes later within 24 hours postop
changes in 1-minute heart rate average from post-intervention to 30 minutes later as assessed using a data collection computer connected to patient's bedside monitor | immediately after each intervention and 30 minutes later within 24 hours postop
changes in 1-minute respiratory rate average from post-intervention to 30 minutes later as assessed using a data collection computer connected to patient's bedside monitor | immediately after each intervention and 30 minutes later within 24 hours postop

CONTACTS AND LOCATIONS:
Overall Officials: Celine Gelinas, PhD, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Bauer BA, Cutshall SM, Wentworth LJ, Engen D, Messner PK, Wood CM, Brekke KM, Kelly RF, Sundt TM 3rd. Effect of massage therapy on pain, anxiety, and tension after cardiac surgery: a randomized study. Complement Ther Clin Pract. 2010 May;16(2):70-5. doi: 10.1016/j.ctcp.2009.06.012. Epub 2009 Jul 14. PMID 20347836
- [Background] Braun LA, Stanguts C, Casanelia L, Spitzer O, Paul E, Vardaxis NJ, Rosenfeldt F. Massage therapy for cardiac surgery patients--a randomized trial. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1453-9, 1459.e1. doi: 10.1016/j.jtcvs.2012.04.027. Epub 2012 Sep 7. PMID 22964355
- [Derived] Boitor M, Martorella G, Laizner AM, Maheu C, Gelinas C. The Effectiveness of Hand Massage on Pain in Critically Ill Patients After Cardiac Surgery: A Randomized Controlled Trial Protocol. JMIR Res Protoc. 2016 Nov 7;5(4):e203. doi: 10.2196/resprot.6277. PMID 27821384